CLINICAL TRIAL: NCT04961372
Title: Socio-psychological Status of Healthcare Workers During SARS-CoV2 Pandemic
Status: Completed | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Hakan Gokalp TAS, Anesthesiology And Reanimation specialist,MD, Erzincan University
Other Study IDs: ErzincanUniversity
Record Dates: First submitted 2021-07-01; First posted 2021-07-14 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Depression, Anxiety
Keywords: Depression; Anxiety; Healthcare Workers
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthcare Workers: All healthcare professionals working at Gümüşhane Şiran Government Hospital
  Interventions: Other: Survey
- Non-Healthcare Workers: Twice the number of health workers included in the study, non-health worker volunteers
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — PHQ9 Depression Scale for evaluating depression, GAD7 Anxiety Score for evaluating anxiety, WSAS Score for evaluating Work and Social Adjustment

SUMMARY:
The aim of our study is to investigate the presence of depression, anxiety and fear in healthcare workers during the SARS-CoV2 pandemic process, to evaluate their work and social life situations, as well as to evaluate the perspectives of the entire population towards hospital admission, surgery decision and vaccination.

DETAILED DESCRIPTION:
Severe Acute Respiratory Syndrome - Corona Virus 2 (SARS-CoV2) was detected by the Chinese Center for Disease Control and Prevention on 7 January 2020 in a patient with atypical pneumonia in Wuhan, China, via a nasopharyngeal swab. On March 11, 2020, the World Health Organization declared it a "Pandemic". SARS-CoV2 quickly turned into a global epidemic, with a total of 134,957,021 confirmed cases and 2,918,752 deaths reported in April 2021.Since SARS-CoV2 is a highly contagious disease, the risk of infection in healthcare workers is quite high. In one of the earliest studies in Wuhan, 29 percent of patients (40 out of 138) were reported to be healthcare workers. A report from the American Centers for Disease Control and Prevention (CDC) stated that a total of 9,282 healthcare workers were diagnosed with COVID-19, including 27 deaths, between February 12 and April 9, 2020. Eleven to nineteen percent of COVID-19 cases have been identified as healthcare professionals.As the investigators have seen in studies of SARS or Ebola outbreaks, the sudden onset of an immediately life-threatening epidemic can place an extraordinary amount of pressure on healthcare workers. Increased workload, physical fatigue, inadequate personal equipment, nosocomial transmission, and having to make ethically difficult decisions can have dramatic effects on their physical and mental health. The weight of working conditions together with the risk of illness of their social environment and families can cause mental health problems such as fear and anxiety in healthcare workers.When an effective vaccination program is in place, population uptake should be as high as possible to achieve herd immunity. Vaccination hesitancy, defined as a delay in acceptance or rejection of vaccination despite the availability of vaccination services, is one of the barriers to this. It is a complex special case that varies with time, place, and vaccines. It is influenced by factors such as peace of mind, convenience, and trust. Vaccine hesitations have been identified as one of the ten global health threats of 2019.The aim of our study is to investigate the presence of depression, anxiety and fear in healthcare workers during the SARS-CoV2 pandemic process, to evaluate their work and social life situations, as well as to evaluate the perspectives of the entire population towards hospital admission, surgery decision and vaccination.

ELIGIBILITY:
Inclusion Criteria:

* All healthcare workers aged between 18-65 who works at Siran Government Hospital

Exclusion Criteria:

* Participants who did not agree to participate in the study
* Uncooperative participants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All healthcare workers aged between 18-65 who works at Siran Government Hospital (111 volunteers) and 222 healthy volunteers who are non-healthcare workers.
Sampling Method: Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 Score | 6 Months
  Depression Score.1-4 Minimal depression,5-9 Mild depression,10-14 Moderate depression,15-19 Moderately severe depression,20-27 Severe depression
Generalised Anxiety Disorder Assessment Score | 6 Months
  Anxiety Score. 0-4: minimal anxiety,5-9: mild anxiety,10-14: moderate anxiety,15-21: severe anxiety
Work and Social Adjustment Score | 6 Months
  Work and Social Adjustment Score. WSAS score above 20 appears to suggest moderately severe or worse psychopathology. Scores between 10 and 20 are associated with significant functional impairment but less severe clinical symptomatology. Scores below 10 appear to be associated with subclinical populations

CONTACTS AND LOCATIONS:
Locations (1):
- Siran Government Hospital, Gümüşhane, Siran, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] WHO. WHO Coronavirus (COVID-19) Dashboard [Web Page]. 2021 [updated 11.04.2021. WHO Coronavirus (COVID-19) Dashboard]. Available from: https://covid19.who.int/.
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] CDC COVID-19 Response Team. Characteristics of Health Care Personnel with COVID-19 - United States, February 12-April 9, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 17;69(15):477-481. doi: 10.15585/mmwr.mm6915e6. PMID 32298247
- [Background] Liu X, Kakade M, Fuller CJ, Fan B, Fang Y, Kong J, Guan Z, Wu P. Depression after exposure to stressful events: lessons learned from the severe acute respiratory syndrome epidemic. Compr Psychiatry. 2012 Jan;53(1):15-23. doi: 10.1016/j.comppsych.2011.02.003. Epub 2011 Apr 12. PMID 21489421
- [Background] Lung FW, Lu YC, Chang YY, Shu BC. Mental Symptoms in Different Health Professionals During the SARS Attack: A Follow-up Study. Psychiatr Q. 2009 Jun;80(2):107-16. doi: 10.1007/s11126-009-9095-5. Epub 2009 Feb 27. PMID 19247834
- [Background] Wu P, Fang Y, Guan Z, Fan B, Kong J, Yao Z, Liu X, Fuller CJ, Susser E, Lu J, Hoven CW. The psychological impact of the SARS epidemic on hospital employees in China: exposure, risk perception, and altruistic acceptance of risk. Can J Psychiatry. 2009 May;54(5):302-11. doi: 10.1177/070674370905400504. PMID 19497162
- [Background] Fontanet A, Cauchemez S. COVID-19 herd immunity: where are we? Nat Rev Immunol. 2020 Oct;20(10):583-584. doi: 10.1038/s41577-020-00451-5. PMID 32908300
- [Background] Ashby B, Best A. Herd immunity. Curr Biol. 2021 Feb 22;31(4):R174-R177. doi: 10.1016/j.cub.2021.01.006. Epub 2021 Jan 12. PMID 33621500
- [Background] Swaminathan S. The WHO's chief scientist on a year of loss and learning. Nature. 2020 Dec;588(7839):583-585. doi: 10.1038/d41586-020-03556-y. No abstract available. PMID 33335314
- [Background] MacDonald NE; SAGE Working Group on Vaccine Hesitancy. Vaccine hesitancy: Definition, scope and determinants. Vaccine. 2015 Aug 14;33(34):4161-4. doi: 10.1016/j.vaccine.2015.04.036. Epub 2015 Apr 17. PMID 25896383
- [Background] Thangaraju P, Venkatesan SJCMJ. WHO Ten threats to global health in 2019: Antimicrobial resistance. 2019;44(3):1150-1.